CLINICAL TRIAL: NCT05000190
Title: Acute and Chronic Effect of 250 mg Citicoline Consumption on Attention in Adults: A Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PEP-2101
Record Dates: First submitted 2021-08-03; First posted 2021-08-11 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Attention
Keywords: cognition; attention; attentional performance; CPT-III; citicoline
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 250 mg citicoline (Experimental): Opaque capsule
  Interventions: Dietary Supplement: Active capsule
- 0 mg citicoline (Placebo Comparator): Opaque capsule matched in appearance to the active capsule
  Interventions: Other: Placebo capsule

INTERVENTIONS:
Dietary Supplement: Active capsule — 1 capsule daily for 28 days
  Arms: 250 mg citicoline
Other: Placebo capsule — 1 capsule daily for 28 days
  Arms: 0 mg citicoline

SUMMARY:
The primary study objectives are to test whether among a sample of healthy adults consuming: (1) a single capsule containing 250 mg citicoline has an effect on attentional performance 1, 2 and 3 h post-dose compared to placebo (acute effect), and (2) capsule containing 250 mg citicoline per day for 28 consecutive days has an effect on attentional performance compared to placebo (chronic effect).

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating females, 18-60 years of age
* Self-report of good health
* Willing to maintain habitual diet, physical activity pattern, and body weight throughout the trial
* Willing to maintain current dietary supplement use (e.g., multi-vitamin or other supplements approved by investigator, stimulants excluded) throughout the 28 days of the trial. On test days, participant agrees not to take any of their usual dietary supplements until dismissal from University of Georgia.
* Willing to abstain from alcohol consumption and avoid vigorous physical activity for 24 h prior to all test visits.
* Absence of health conditions that would prevent fulfillment of study requirements as judged by the Investigator on the basis of medical history.
* Understanding the study procedures and willing to provide informed consent to participate in the study and authorization to release relevant protected health information to the study investigator.

Exclusion Criteria:

* Failure to meet any one of the inclusion criteria
* Potential participant will be excluded if the individual is being paid to do work by Dr. O'Connor, is unwilling to comply with safety instructions (e.g., to wear a face covering) or reports:
* Vision problems that cannot be corrected with glasses or contact lenses
* usual daily consumption of ≥ 500 mg caffeine
* Consumption of caffeine or other stimulants, such as stimulant medication commonly used for ADHD (e.g. Ritalin or Adderall), within 12 h of testing. Prescription medications are allowed as long as they do not interfere with testing.
* Major trauma or major surgical event within 6 months of screening
* Known intolerance, sensitivity or allergy to any ingredients in the study products
* Extreme dietary habits, as judged by the Investigator
* Moderate or higher intensity exercise of 15 or more minutes completed fewer than 3-h prior to a laboratory testing session.
* Consumption of food or caloric drinks fewer than 2-h prior to the laboratory testing session.
* Consumption of supplements, vitamins and multi-vitamins prior to testing on testing days. Participants can take dietary supplements that they have agreed to maintain on testing days after completing the testing visit.
* Any history of a diagnosed psychiatric or neurobehavioral (e.g., ADHD) disorder
* A history of frequent gastrointestinal distress in response to meals or medicine
* History of cancer in the prior two years, except for non-melanoma skin cancer
* Recent history (within 12 months of screening) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as > 14 drinks per week (1 drink=12 oz beer, 5 oz wine, or 1.5 oz distilled spirits).
* Exposure to citicoline within 30 d prior to screening
* Participant has a condition the investigator believes would interfere with his/her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk
* Increased risk of exposure to COVID-19
* Increased risk of a severe reaction to exposure to COVID-19
* Participation in a PepsiCo study at the University of Georgia for at least 6 months from signing the consent form
* Participation in any clinical trial for at least 30 days from signing the consent form

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
Errors of commission after 28-day consumption (chronic effect) | Post treatment Day 29 minus pre-treatment (baseline Day 1) change scores
  Attention performance during the Connors Continuous Performance Test- version III (CPT-III)

SECONDARY OUTCOMES:
Errors of commission after acute dosing (single dose on Day 1, the first of 28 daily doses) | Change from pre-dose baseline to 1 hour, 2 hours and 3 hours post dose (baseline Day 1)
  Attention performance during the (CPT)-III
Errors of omission after acute dosing | Change from pre-dose baseline to 1 hour, 2 hours and 3 hours post dose (baseline Day 1)
  Attention performance during the CPT-III
Errors of omission after chronic dosing | Post treatment Day 29 minus pre-treatment (baseline Day 1) change scores
  Attention performance during the CPT-III
Reaction time after acute dosing | Change from pre-dose baseline to 1 hour, 2 hours and 3 hours post dose (baseline Day 1)
  Attention performance indicator from the CPT-III
Reaction time after chronic dosing | Post treatment Day 29 minus pre-treatment (baseline Day 1) change scores
  Attention performance indicator from the CPT-III
For the acute study only, expectation for change in mental task performance associated with consuming one capsule that may contain citicoline | Immediately post-dose (baseline Day 1)
  Measured by two item questionnaire, 5 selections each item, from very much worse to very much better than expected mental task performance if assigned to active and if assigned to placebo
For acute study only, sleep behavior the night prior to testing | Upon arrival (baseline Day 1)
  Questionnaire about number of hours of sleep last night
For the acute study only, motivation to complete the attention task | Change from pre-dose baseline to 1 hour, 2 hours and 3 hours post dose immediately prior to tests of attention
  Single question, How do you feel right now, rated on visual analog scale (VAS) from 0 (no motivation at all) to 100 (strongest degree of motivation imaginable)
For the acute study only, feelings of mental energy and fatigue | Immediately prior to the test of attention, change from pre-dose baseline to 1 hour, 2 hours and 3 hours post dose
  6 questions rated by visual analog scale (VAS) from 0 mm (weakest) to 100 mm (strongest) feelings
For the acute study only, mood states (anxiety) | Immediately prior to the test of attention, change from pre-dose baseline to 1 hour, 2 hours and 3 hours post dose mood states, immediately prior to tests of attention
  Profile of Mood States (POMS) questionnaire, 30 questions, How do you feel right now, rated 0 (not at all) to 4 (extremely)
For the acute study only, high frequency (HF) and low frequency (LF) domains of heart rate variability, a biomarker of cognitive function, during the tests of attention | Change from pre-dose baseline to 1 hour, 2 hours and 3 hours post dose
  Beats per minute via wearable heart rate monitor
For the chronic study only, expectation for change in mental task performance associated with consuming one capsule daily for 28-days that may contain citicoline | Change from post-dose baseline Day 1 to Day 29 measured by
  Two item questionnaire, 5 selections each item, from very much worse to very much better than expected mental task performance if had been assigned to active and if had been assigned to placebo for 28 days
For the chronic study only, sleep behavior the night prior to testing | Change from number of hours of sleep the night before baseline Day 1 versus the number of hours of sleep the night before Day 29
  Questionnaire about number of hours of sleep last night
For the chronic study only, motivation to complete the attention task | Change from pre-dose baseline Day 1 to Day 29
  Single question, How do you feel right now, rated on visual analog scale (VAS) from 0 (no motivation at all) to 100 (strongest degree of motivation imaginable)
For the chronic study only, feelings of mental energy and fatigue | Immediately prior to test of attention, change from pre-dose baseline Day 1 to Day 29
  6 questions rated by visual analog scale (VAS) from 0 mm (weakest) to 100 mm (strongest) feelings
For the chronic study only, mood states (anxiety) questionnaire | Immediately prior to test of attention, change from pre-dose baseline Day 1 to Day 29
  Profile of Mood States (POMS) questionnaire, , 30 questions, How do you feel right now, rated 0 (not at all) to 4 (extremely)
For the chronic study only, high frequency (HF) and low frequency (LF) domains of heart rate variability, a biomarker of cognitive function, during the tests of attention | Change from pre-dose baseline Day 1 to Day 29
  Beats per minute via wearable heart rate monitor

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J O'Connor, PhD, Principal Investigator — University of Georgia, Athens
Locations (1):
- University of Georgia, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: No